CLINICAL TRIAL: NCT05461989
Title: Physical Activity Barriers in Adolescent Hypertension Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, E.Burcu ÖZCAN, Physiotherapist (MSc), Hacettepe University
Other Study IDs: GO 22/505
Record Dates: First submitted 2022-07-09; First posted 2022-07-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior | interventions — Hand Strength; Vascular Stiffness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- primary hypertension: adolesence primary hypertension patients
  Interventions: Other: Anthropometric measurement; Other: Level of Physical Activity; Other: Physical Activity Barriers Scale; Other: Hand Grip Strength; Other: Arterial stiffness
- secondary hypertension: adolesence secondary hypertension patients
  Interventions: Other: Anthropometric measurement; Other: Level of Physical Activity; Other: Physical Activity Barriers Scale; Other: Hand Grip Strength; Other: Arterial stiffness

INTERVENTIONS:
Other: Anthropometric measurement — It will be measured with the Xiaomi Body Composition Scale II, and a total of 9 measurements will be made as a result of the measurements.
Other: Level of Physical Activity — The scale to be used for this purpose is the Child Physical Activity Questionnaire (CPAQ) developed by Kowalski et al. It is a seven-day self-reported recall scale designed to assess moderate-intensity physical activity in children aged 8-14 years. CFAQ is designed to be implemented throughout the school year.
Other: Physical Activity Barriers Scale — It consists of three surveys in total, which are:
  A) Scale of Expectations Regarding Physical Activity for Children
  B) Children's perception of family support regarding physical activity scale
  C) Physical Activity Barriers Scale for Parents
Other: Hand Grip Strength — Hand grip strength will be measured using a hand dynamometer (Jamar, Sammons Preston, Rolyon, Bolingbrook, IL).
Other: Arterial stiffness — Arterial stiffness will be evaluated using the pulse wave velocity (PWV) technique with the blood pressure holter-ABPM (Mobil-O-Graph, I.E.M., Stolberg, Germany) device. The measurement is made from the non-dominant arm based on the principle of blood pressure measurement with the appropriate cuff determined according to the arm diameter. After two consecutive measurements taken 30 seconds apart, the average of the measurement values will be recorded.

SUMMARY:
One of the most prevalent chronic disorders in children, especially teenagers, is hypertension . The prevalence of hypertension has significantly increased in recent years, particularly with the rise in obesity. It has been demonstrated that hypertension is a significant, controllable risk factor for cardiovascular disease and that it is linked to atherosclerosis in children. Additionally, in patients with hypertension who were monitored from infancy to adulthood, it was discovered that the unfavorable cardiac alterations and vascular damage linked to hypertension were linked to early cardiovascular disease in adults. Therefore, the key to preventing cardiovascular disease in children and adolescents-especially when risk factors like obesity, diabetes, or chronic renal disease are present-is early diagnosis and effective treatment of hypertension. Insufficient exercise and sedentary lifestyles are additional risk factors for pediatric hypertension.Investigating physical activity barrier in teenage hypertension patients is vital in light of all these factors as well as studies on adolescents' inadequate physical activity. The literature is lacking studies examining the obstacles to physical exercise faced by people with adolescent hypertension, hence this topic is open for investigation.

DETAILED DESCRIPTION:
One of the most prevalent chronic disorders in children, especially teenagers, is hypertension . The prevalence of hypertension has significantly increased in recent years, particularly with the rise in obesity . Primary hypertension, also known as essential hypertension, which was once thought to be an adult condition, is becoming more prevalent in the pediatric population, partly because of the obesity pandemic . Children who are obese have a three times higher risk of developing hypertension than children who are not obese . Based on the etiology, hypertension can be divided into two types: primary or essential hypertension, which has no known cause, and secondary hypertension, which has a known cause. Stage I (mild) hypertension is the most common symptom of primary hypertension, which is also linked to a favorable family history . Very young children, those with stage II hypertension, and those with clinical signs suggesting systemic disorders linked to hypertension should all be evaluated for secondary hypertension. An underlying vascular, neurological, endocrine, or renal parenchymal illness may cause secondary hypertension .

It has been demonstrated that hypertension is a significant, controllable risk factor for cardiovascular disease and that it is linked to atherosclerosis in children. Additionally, in patients with hypertension who were monitored from infancy to adulthood, it was discovered that the unfavorable cardiac alterations and vascular damage linked to hypertension were linked to early cardiovascular disease in adults.Therefore, the key to preventing cardiovascular disease in children and adolescents-especially when risk factors like obesity, diabetes, or chronic renal disease are present-is early diagnosis and effective treatment of hypertension.

Insufficient exercise and sedentary lifestyles are additional risk factors for pediatric hypertension. Low levels of physical activity and hypertension have a continuous, temporal, and independent association, according to epidemiological research . According to data, 80% of kids and teenagers in 105 countries do not engage in the recommended amount of physical exercise, which is at least 60 minutes of moderate to strenuous activity per day.Additionally, many kids and teenagers engage in sedentary activities for more than 4 hours per day, even though less than 2 hours per day are advised for screen-based entertainment (such as watching TV, using a computer, and playing video games). According to research, children and adolescents who watch television or spend too much time on screens had lower fitness levels, worse self-esteem, less prosocial behavior, and higher systolic and diastolic blood pressure. Prospective research regularly demonstrates that exercise shields adults from high blood pressure. Physical activity has been dubbed a "poly-drug" for its preventive and therapeutic effects in reducing the global health burden of cardiovascular disease, increasing physiological function, and slowing cardiovascular aging.Investigating physical activity barrier in teenage hypertension patients is vital in light of all these factors as well as studies on adolescents' inadequate physical activity. The literature is lacking studies examining the obstacles to physical exercise faced by people with adolescent hypertension, hence this topic is open for investigation.

ELIGIBILITY:
For Primary Hypertension

Inclusion Criteria:

* Being 10-19 years old,
* Being diagnosed with primary hypertension,
* Being clinically stable and no drug/drug dose changes for the last four weeks,
* Determined to be voluntary to participate in the study

Exclusion Criteria:

* Having a neurological, cognitive or orthopedic disease that will affect the measurements,
* Severe respiratory system disease (FEV1 <35%; FVC <50%),
* Having acute infection,
* Having malignancy,
* Receiving hormone replacement therapy,
* Body mass index >40 kg/m²,
* Ejection fraction less than 50%,
* Having uncontrolled hypertension,
* Individuals with diabetes will not be included in the study.

For Secondary Hypertension

Inclusion Criteria:

* Being 10-19 years old,
* Being diagnosed with secondary hypertension,
* Being clinically stable and no drug/drug dose changes for the last four weeks,
* Not being under high-dose glucocorticoid therapy (2 mg/kg/day),
* Not taking intravenous biologic or conventional immunosuppressive therapy (including pulsed steroids) in the past month
* Determined to be voluntary to participate in the study

Exclusion Criteria:

* Having a neurological, cognitive or orthopedic disease that will affect the measurements,
* Severe respiratory system disease (FEV1 <35%; FVC <50%),
* Having acute infection,
* Having malignancy,
* Receiving hormone replacement therapy,
* Body mass index >40 kg/m²,
* Ejection fraction less than 50%,
* Having uncontrolled hypertension,
* Individuals with diabetes will not be included in the study.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescent primary and secondary hypertension patients
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
physical activity barriers | 12 months
  With a scale consisting of three questionnaires in total (Parent Physical Activity Barriers scale, the Child Physical Activity Outcome Expectancies Scale, and the Child Physical Activity Home Environment scale), the barriers of individuals to physical activity will be evaluated. As a result of these evaluations, it will guide us to understand the causes of physical activity barriers in primary and secondary hypertension patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No